CLINICAL TRIAL: NCT05035875
Title: Evaluation of Diaphragm in Chronic Obstructive Pulmonary Disease Patients Using Ultrasonography in Relation to Disease Severity in Fayoum University Hospital
Brief Title: Evaluation of Diaphragm in Chronic Obstructive Pulmonary Disease Patients by Ultrasound in Relation to Severity
Status: Completed | Type: Observational
Sponsor: Enas Sayed Farhat (Other)
Responsible Party: Sponsor-Investigator, Enas Sayed Farhat, fayoum university hospital, Fayoum University Hospital
Organization: Fayoum University Hospital (Other)
Other Study IDs: M 448
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: ultrasonography, diaphragm, COPD, Fayoum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 40 COPD patients: all participants were subjected to : history - clinical examination - spirometry - ultrasound evaluation of diaphragmatic function
  Interventions: Device: ultrasonography
- 40 healthy individuals: all participants were subjected to : history - clinical examination - spirometry - ultrasound evaluation of diaphragmatic function
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — ultrasound assessment of diaphragm function

SUMMARY:
The study of the diaphragm is an important point in the assessment of COPD patients.

Ultrasonographic evaluation of the diaphragm is considered a simple, non-invasive, available bedside technique. Ultrasonography can be used for evaluation of the site, structure, and motion of the diaphragm, assessment of excursion, and thickness.

The aim of the study is ultrasonographic assessment of the diaphragm in COPD patients and its relation to disease severity

DETAILED DESCRIPTION:
The study was conducted on eighty patients, forty COPD patients who were diagnosed and classified into four groups according as following: The first group: included 10 patients with a mild stage. The second group: included 10 patients with a moderate stage. The third group: included 10 patients with a severe stage. The fourth group: included 10 patients with a very severe stage. The study also included forty healthy individuals of the same age and sex as COPD patients. All participants gave their informed consent for inclusion before sharing in the study. Every person was submitted to: Full medical history, Clinical examination,Chest x-ray, spirometry and ultrasonographic assessment of diaphragm function (thickness and excursion)

ELIGIBILITY:
Inclusion Criteria:

* • Stable COPD patients aged more than 40 years who were diagnosed and classified into four groups of severity according to GOLD 2020.

  * Age and sex-matched healthy controls

Exclusion Criteria:

* • Patient with a known neuromuscular disorder.

  * Patient with known anatomical malformation of the diaphragm.
  * Post abdominal or thoracic surgery.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 COPD patients and 40 age matched healthy control
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
measure diaphragmatic thickness by ultrasound | 1 year study
  measure diaphragmatic thickness at total lung capacity and residual volume in millimetres to calculate diaphragm thickness fraction
measure diaphragm excursion by ultrasound | 1 year study
  measure diaphragm excursion in centimetres at zone of apposition

SECONDARY OUTCOMES:
spirometry assessment | 1 year study
  value of forced expiratory volume in first second is assessed as a percentage of normal by spirometry to assess disease severity
questionnaires | 1 year study
  ( modified medical research council and chronic obstructive pulmonary disease assessment test) to detect severity of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Enas S Farhat, MD, Principal Investigator — Fayoum University Hospital
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
after the submission is finished, the individual participant data will be shared to other researchers